CLINICAL TRIAL: NCT00443664
Title: External Micropulse Diode Laser Transscleral Trabeculoplasty(EMDLT) For Severe Open Angle Glaucoma
Brief Title: External Micropulse Diode Laser Transscleral Trabeculoplasty (EMDLT) for Severe Open Angle Glaucoma
Acronym: EMDLT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Paul TK Chew, MBBS,MMedoph, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB-A/06/165
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EXTERNAL MICROPULSE DIODE LASER TRANSSCLERAL TRABECULOPLASTY

SUMMARY:
To prove that external contact micropulse diode laser trabeculoplasty (EMDLT) can significantly lower intraocular pressure in cases of advanced open angle glaucoma.

DETAILED DESCRIPTION:
Micropulse diode laser trabeculoplasty applied through a gonioscopy len has been shown to be effective in lower the pressure for patients with primary open angle glaucoma (POAG). We believe that applied externally, the contact diode micropulse laser will be effective in lowering intraocular pressure for patients with advance open angle glaucoma with minimal side effects

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of Primary Open Angle Glaucoma

  * Advanced glaucoma with intraocular pressure higher than 21mmHg on one or more topical medications (for at least 2 months)
  * Visual acuity worse than 6/6
  * Age more than 21 years
  * Poor candidate for additional filtration surgery

Exclusion Criteria:

* • Age less than 21 years

  * Any eye surgery within 2 months of enrolment
  * Any patient with rubeosis
  * Unable to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-06; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The amount of pressure lowering after EXTERNAL MICROPULSE DIODE LASER TRANSSCLERAL TRABECULOPLASTY (EMDLT) treatment.

SECONDARY OUTCOMES:
Study of safety of EXTERNAL MICROPULSE DIODE LASER TRANSSCLERAL TRABECULOPLASTY (EMDLT) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul TK Chew, MBBS,MMedOph, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] The Glaucoma Laser Trial (GLT). 2. Results of argon laser trabeculoplasty versus topical medicines. The Glaucoma Laser Trial Research Group. Ophthalmology. 1990 Nov;97(11):1403-13. PMID 2255512
- [Background] Kramer TR, Noecker RJ. Comparison of the morphologic changes after selective laser trabeculoplasty and argon laser trabeculoplasty in human eye bank eyes. Ophthalmology. 2001 Apr;108(4):773-9. doi: 10.1016/s0161-6420(00)00660-6. PMID 11297496
- [Background] Ho CL Micropulse Diode Trans-scleral Cyclophotocoagulation Asian Journal of ophth. 2001 supplement. vol 3,no 3,4
- [Background] Ingvoldstad DD, Krishna R, Willoughby L. MicroPulse Diode Laser Trabeculoplasty versus Argon Laser Trabeculoplasty in the treatment of Open angle glaucoma. Presented at ARVO 2005, Poster 123.